CLINICAL TRIAL: NCT00856115
Title: Appraisal Delay and Disparities in Timely Cancer Diagnosis
Brief Title: Differences in Timely Cancer Diagnosis in African American and Caucasian Patients With Newly Diagnosed Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE4208; P30CA043703 (NIH); CASE4208 (Other: Case Comprehensive Cancer Center); CASE 4208-CC498 (Other: Cancer Center IRB)
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Colorectal Cancer
Keywords: stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- African American Female
  Interventions: Other: medical chart review; Other: questionnaire administration; Other: study of socioeconomic and demographic variables; Other: survey administration
- African American Male
  Interventions: Other: medical chart review; Other: questionnaire administration; Other: study of socioeconomic and demographic variables; Other: survey administration
- Caucasian Female
  Interventions: Other: medical chart review; Other: questionnaire administration; Other: study of socioeconomic and demographic variables; Other: survey administration
- Caucasian Male
  Interventions: Other: medical chart review; Other: questionnaire administration; Other: study of socioeconomic and demographic variables; Other: survey administration

INTERVENTIONS:
Other: medical chart review — Patient charts are reviewed to obtain medical data.
Other: questionnaire administration — Patients undergo a 45-60 minute interview to obtain information on variations in symptom perception, assessment, and patient-physician communication process. Patients are assessed by sociodemographic characteristics (i.e, education, gender, age, insurance status, employment status, income, race/ethnicity, and religiosity), information of close confidants (i.e., relationship, family history of cancer, and caregiver/decision-making status), and physician characteristics. Patients are also assessed by the Trust in the Health Care System, DMPQ, RCS, Brief COPE scale, Lukwago Religiosity scale, and RAND Social Support Survey questionnaires.
Other: study of socioeconomic and demographic variables — Patients are assessed by sociodemographic characteristics (i.e, education, gender, age, insurance status, employment status, income, race/ethnicity, and religiosity).
Other: survey administration — Patients are also assessed by the Trust in the Health Care System, DMPQ, RCS, Brief COPE scale, Lukwago Religiosity scale, and RAND Social Support Survey questionnaires.

SUMMARY:
RATIONALE: Gathering information about timely diagnosis in African American and Caucasian patients with newly diagnosed colorectal cancer may help doctors learn more about factors that influence a diagnosis and plan the best treatment.

PURPOSE: This phase I trial is studying differences in timely cancer diagnosis in African American patients and in Caucasian patients with newly diagnosed colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify and examine the factors that influence appraisal and diagnostic delay by focusing on recognition, perception, communication, and response to pre-diagnosis cancer symptoms in African American and Caucasian patients with newly diagnosed colorectal cancer.

OUTLINE: This is a multicenter study. Patients are stratified according to race (African-American vs Caucasian) and gender (male vs female).

Patients undergo a 45-60 minute interview to obtain information on variations in symptom perception, assessment, and patient-physician communication process. Patients are assessed by sociodemographic characteristics (i.e, education, gender, age, insurance status, employment status, income, race/ethnicity, and religiosity), information of close confidants (i.e., relationship, family history of cancer, and caregiver/decision-making status), and physician characteristics. Patients are also assessed by the Trust in the Health Care System, DMPQ, RCS, Brief COPE scale, Lukwago Religiosity scale, and RAND Social Support Survey questionnaires.

Patient charts are reviewed to obtain medical data.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older
* Cognitively able to participate in an interview
* Diagnosed with Colorectal cancer
* Patient at University Hospitals, Case Western Reserve University, or Cleveland Clinic Foundation
* diagnosed within 6 months of the scheduled interview
* have no prior history of colon cancer or cancer of any other major organ system
* any stage of cancer
* Patient will have described their symptoms to their PCPs
* Patient will have acted as their own decision maker
* Must be African American or Caucasian

Exclusion Criteria

* No disease discovered by previous routine screening or by other unintentional detection procedure (i.e., without symptom appraisal process or communicating specific symptoms to physicians)
* Not living in nursing or assisted living facilities
* Cognitive impairment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: African American patients and Caucasian patients with newly diagnosed colorectal cancer.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2008-11; Primary Completion 2010-10 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Factors that influence appraisal and diagnostic delay | 45-60 minute interview

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Harris-Haywood, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (4):
- United States (4):
  - Lake/University Ireland Cancer Center, Cleveland, Ohio
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Southwest General Health Center, Cleveland, Ohio
  - UH-Green Road, South Euclid, Ohio